CLINICAL TRIAL: NCT02395393
Title: Confocal Fluorescence Microscopy of the Human Airways in Diagnostics of Lung Transplantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is planned for later
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Levent Midyat, MD, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-P00017377
Record Dates: First submitted 2015-03-10; First posted 2015-03-23 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Disorder Related to Lung Transplantation
Keywords: Acute rejection; Chronic rejection; Confocal microscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung transplant recipients (Other): In patients scheduled for bronchoscopy as part of regular clinical care/diagnostic workup, the investigators will offer the patient concurrent confocal microscopy imaging to be performed during the bronchoscopic procedure. A 1.4mm or 1.9mm diameter Alveoflex Confocal MiniprobeTM (MaunaKea Technologies, France) will be deployed down the working channel of the standard bronchoscope and advanced distally into the alveoli.
  Interventions: Device: Alveoflex Confocal MiniprobeTM

INTERVENTIONS:
Device: Alveoflex Confocal MiniprobeTM — -Alveolar imaging

SUMMARY:
Bronchoscopy-guided tissue sampling is a central technique in many diseases including diagnosing and staging lung cancers, diagnosing interstitial lung diseases, and acute and/or chronic rejections following lung transplantation. Confocal fluorescence microscopy is a novel technique used for real-time microscopic imaging of proximal and distal airways, microvessels, and inflammatory cells. We hypothesize that confocal fluorescence microscopy images of airways and alveolar structures during standard bronchoscopy could help recognize and classify the presence or absence of acute or chronic rejection in lung transplant recipients.

DETAILED DESCRIPTION:
Bronchoscopy-guided tissue sampling is a central technique in many diseases including diagnosing and staging lung cancers, diagnosing interstitial lung diseases, and acute and/or chronic rejections following lung transplantation. Confocal fluorescence microscopy is a novel technique used for in vivo microscopic imaging of proximal and distal airways including bronchial and alveolar walls, microvessels, and inflammatory cells. We hypothesize that confocal fluorescence microscopy images of bronchiolar and alveolar structures during standard bronchoscopy could help recognize and classify the presence or absence of acute or chronic rejection in lung transplant recipients.

The objectives and outcomes of this study are:

1. To assess the safety of confocal microscopy imaging in pediatric patients
2. To create diagnostic criteria for fibered confocal fluorescence microscopy image interpretation of acute and chronic rejections following lung transplantation
3. To determine the sensitivity and specificity of confocal imaging in these patient groups compared to the transbronchial biopsies
4. Correlate confocal images to FEV1 results
5. Correlate with CXRs and/or CT images

ELIGIBILITY:
Inclusion Criteria:

* to be older than six years of age
* to be undergoing surveillance or clinically indicated bronchoscopies with transbronchial biopsy as part of their routine care
* to be willing and able to comply with study procedures and provide written informed consent/assent to participate in the study

Exclusion Criteria:

* to be unwilling to consent
* to be unable to safely tolerate a bronchoscopic procedure
* to have any contraindications to short-acting anesthetic agents
* to have any contraindications to transbronchial biopsies

Ages: 6 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of confocal imaging in these patient groups compared to the transbronchial biopsies | One year
  Correlate confocal images to histolopathologic findings of acute rejection, chronic rejection, and no evidence of rejection

SECONDARY OUTCOMES:
Number of participants with adverse events | One year
  Monitor for serious adverse events
Correlation of confocal images with FEV1 results | One year
  Measure the degree of fibrosis/collagen by confocal imaging and compare to FEV1 values

CONTACTS AND LOCATIONS:
Overall Officials: Gary Visner, DO, Study Director — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Izbicki G, Shitrit D, Yarmolovsky A, Bendayan D, Miller G, Fink G, Mazar A, Kramer MR. Is routine chest radiography after transbronchial biopsy necessary?: A prospective study of 350 cases. Chest. 2006 Jun;129(6):1561-4. doi: 10.1378/chest.129.6.1561. PMID 16778275
- [Background] Hanson RR, Zavala DC, Rhodes ML, Keim LW, Smith JD. Transbronchial biopsy via flexible fiberoptic bronchoscope; results in 164 patients. Am Rev Respir Dis. 1976 Jul;114(1):67-72. doi: 10.1164/arrd.1976.114.1.67. PMID 937843
- [Background] Thiberville L, Salaun M, Lachkar S, Dominique S, Moreno-Swirc S, Vever-Bizet C, Bourg-Heckly G. Human in vivo fluorescence microimaging of the alveolar ducts and sacs during bronchoscopy. Eur Respir J. 2009 May;33(5):974-85. doi: 10.1183/09031936.00083708. Epub 2009 Feb 12. PMID 19213792
- [Background] Yserbyt J, Dooms C, Decramer M, Verleden GM. Probe-based confocal laser endomicroscopy of the respiratory tract: a data consistency analysis. Respir Med. 2013 Aug;107(8):1234-40. doi: 10.1016/j.rmed.2013.04.018. Epub 2013 May 23. PMID 23706778
- [Background] Thiberville L, Salaun M, Lachkar S, Dominique S, Moreno-Swirc S, Vever-Bizet C, Bourg-Heckly G. Confocal fluorescence endomicroscopy of the human airways. Proc Am Thorac Soc. 2009 Aug 15;6(5):444-9. doi: 10.1513/pats.200902-009AW. PMID 19687217